CLINICAL TRIAL: NCT01754818
Title: Phase 1 Randomized, Double-blind, Placebo-controlled Study of The Safety, Tolerability and Pharmacokinetics of Single, Ascending Oral Doses Of Bendavia in Healthy Volunteers
Brief Title: A Phase 1 Study Examining the Pharmacokinetics and Tolerability of a Single Oral Dose of Bendavia (MTP-131)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SPIO-101
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Pharmacokinetics; volunteers
MeSH Terms: interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo, oral capsule, no active study drug, single dose
  Interventions: Drug: Placebo
- Bendavia 10mg (Experimental): Bendavia, oral capsule, 10mg, single dose
  Interventions: Drug: Bendavia 10mg; Drug: Placebo
- Bendavia 50mg (Experimental): Bendavia, oral capsule, 50mg, single dose
  Interventions: Drug: Bendavia 50mg; Drug: Placebo
- Bendavia 100mg (Experimental): Bendavia, oral capsule, 100mg, single dose
  Interventions: Drug: Bendavia 100mg; Drug: Placebo

INTERVENTIONS:
Drug: Bendavia 10mg
  Arms: Bendavia 10mg
Drug: Bendavia 50mg
  Arms: Bendavia 50mg
Drug: Bendavia 100mg
  Arms: Bendavia 100mg
Drug: Placebo

SUMMARY:
The purpose of this study is to assess the study medication blood levels after administration of a single oral capsule of Bendavia at one of three dose levels. The effects of Bendavia on the volunteers will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females aged between 18 and 65 years of age with signed informed consent.
* Women who are not post-menopausal (without menstrual bleed for >24 months) or surgically sterile must have a negative serum pregnancy test at screening and within 24 hours of treatment with understanding (through informed consent process) to not become pregnant over the duration of the study and must agree to employ an effective form of birth control for the duration of the study.
* Acceptable forms of birth control are: double-barrier contraceptives (condom, diaphragm with spermicide) or intra-uterine device 1 week prior to and at least 30 days post treatment even if hormonal contraceptives are used.

Exclusion Criteria:

* Serum sodium level below the lower limit of the site's clinical laboratory normal range at the study qualification visit,
* Clinically significant laboratory abnormalities as determined by the Principal Investigator at laboratory screening
* Creatinine clearance calculated by the Cockcroft and Gault method calculated to be <90 mL/min for males and <80 mL/min for females
* Clinically significant abnormalities on physical examination,
* Body weight less than 60 or greater than 80 kg and a body mass index of less than 18 kg/m2 or greater than 32 kg/m2,
* Any disease or condition that might compromise the cardiovascular, hematological, renal, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous, or gastrointestinal (including an ulcer) systems,
* History of seizures or history of epilepsy,
* History of serious (Principal Investigator judgment) mental illness,
* Participant in any research involving investigational product within 30 days before planned date of drug administration,
* Positive serology for human immunodeficiency virus type 1 or 2, hepatitis B surface antigen, or hepatitis C,
* Fever greater than 37.5°C at the time of planned dosing,
* Suspicion, or recent history, of alcohol or substance abuse,
* Donated blood or blood products within the past 30 days,
* Women who are pregnant or breastfeeding,
* Employee or family member of the investigational site,
* Subjects who currently smoke cigarettes, cigars, pipes or chew tobacco products or who have used any tobacco product in the 30 days prior to screening,
* Subjects who are either unwilling to agree to refrain from use or found to be using:
* Alcohol, caffeine, xanthine-containing food or beverages, nicotine products and over-the-counter medications with the exception of Tylenol from 24 hours prior to dosing and throughout the confinement period
* Prescription medications from 14 days prior to, and 7 days post, dose (excluding hormonal contraceptives)
* Hormonal contraceptives without concomitant use of double-barrier contraceptives (condom, diaphragm with spermicide) for a period of 7 days prior to, and 30 days post, dose
* Subjects having previous exposure to Bendavia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Mean peak plasma concentration (Cmax) of Bendavia (ng/ml) in each cohort. | Immediately prior to dosing (0hr) to 48 hours post-dose
  Blood drawn at pre-dose (immediately prior to study drug ingestion), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose will be assessed for Bendavia plasma concentrations. Mean Cmax is defined as the mean of maximum concentration reported for each subject by cohort.
Mean Area Under the Curve (AUC) for Bendavia (hr.ng/ml) in the time from dosing to final plasma sample in each cohort. | Immediately prior to dosing (0hr) to 48 hours post-dose
  Blood drawn at pre-dose (immediately prior to study drug ingestion), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose will be assessed for Bendavia plasma concentrations. AUC (0-last) will be calculated using validated pharmacokinetic analysis software and mean AUC for Bendavia is defined as the mean of AUC (0-last) reported for each subject by cohort.
Mean Time post-dose of the peak plasma concentration (Tmax) of Bendavia (hours) in each cohort. | Immediately prior to dosing (0hr) to 48 hours post-dose
  Blood drawn at pre-dose (immediately prior to study drug ingestion), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose will be assessed for Bendavia plasma concentrations. Mean Tmax is defined as the mean of time to reach maximum plasma concentration reported for each subject by cohort.
Mean apparent clearance (CL/F) of Bendavia (ml/hr/kg) in each cohort. | Immediately prior to dosing (0hr) to 48 hours post-dose
  Blood drawn at pre-dose (immediately prior to study drug ingestion), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose will be assessed for Bendavia plasma concentrations. CL/F will be calculated using validated pharmacokinetic analysis software and mean CL/F for Bendavia is defined as the mean of CL/F reported for each subject by cohort.
Mean Volume of Distribution (Vd/F) of Bendavia (ml/kg) in each cohort. | Immediately prior to dosing (0hr) to 48 hours post-dose
  Blood drawn at pre-dose (immediately prior to study drug ingestion), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose will be assessed for Bendavia plasma concentrations. Vd/F will be calculated using validated pharmacokinetic analysis software and mean Vd/F for Bendavia is defined as the mean of Vd/F reported for each subject by cohort.
Mean Half Life(t1/2) of Bendavia (hours) in each cohort. | Immediately prior to dosing (0hr) to 48 hours post-dose
  Blood drawn at pre-dose (immediately prior to study drug ingestion), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose will be assessed for Bendavia plasma concentrations. t1/2 will be calculated using validated pharmacokinetic analysis software and mean t1/2 for Bendavia is defined as the mean of t1/2 reported for each subject by cohort.

SECONDARY OUTCOMES:
Mean Area Under the Curve (AUC) for Bendavia metabolite M1 (hr.ng/ml) in the time from dosing to final plasma sample in each cohort. | Immediately prior to dosing (0hr) to 48 hours post-dose
  Blood drawn at pre-dose (immediately prior to study drug ingestion), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose will be assessed for Bendavia metabolite M1 plasma concentrations. AUC (0-last) will be calculated using validated pharmacokinetic analysis software and mean AUC for Bendavia metabolite M1 is defined as the mean of AUC (0-last) reported for each subject by cohort.
Mean Area Under the Curve (AUC) for Bendavia metabolite M2 (hr.ng/ml) in the time from dosing to final plasma sample in each cohort. | Immediately prior to dosing (0hr) to 48 hours post-dose
  Blood drawn at pre-dose (immediately prior to study drug ingestion), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose will be assessed for Bendavia metabolite M2 plasma concentrations. AUC (0-last) will be calculated using validated pharmacokinetic analysis software and mean AUC for Bendavia metabolite M2 is defined as the mean of AUC (0-last) reported for each subject by cohort.
Mean change in concentration of urinary 8-isoprostane (pg/mg creatinine) from pre-dose through to 48 hours post-dose for each cohort. | Prior to dosing (0hr) to 48 hours post-dose
  Spot urine samples will be collected at pre-dose, 12, 24 and 48 hours post-dose for assay of 8-isoprostane (8-EPIPGF2a) and creatinine. Change from baseline value at each time point assessed will be calculated for each subject. Mean change from baseline is defined as the mean of the change in 8-EPIPGF2a/creatinine for each subject by cohort.
Mean change in concentration of urinary 8-hydroxy-2-deoxyguanosine (ng/mg creatinine) from pre-dose through to 48 hours post-dose for each cohort. | Prior to dosing (0hr) to 48 hours post-dose
  Spot urine samples will be collected at pre-dose, 12, 24 and 48 hours post-dose for assay of 8- hydroxy-2-deoxyguanosine (8-OHDG) and creatinine. Change from baseline value at each time point assessed will be calculated for each subject. Mean change from baseline is defined as the mean of the change in 8-OHDG/creatinine for each subject by cohort.
Number of adverse events observed with and without Bendavia | From time of study drug administration to End of Study (Day 3)
  Adverse events will be tabulated by treatment group. No statistical analysis will be performed.
Mean change from baseline in High Sensitivity C-Reactive Protein (hs-CRP; ng/L) through 48 hours post-dose. | Pre-dose to 48 hours post-dose
  hs-CRP will be evaluated prior to (Baseline) and after (12, 24 and 48 hours) study drug administration. Change from baseline value at each time point assessed will be calculated for each subject. Mean change from baseline is defined as the mean of the change in hs-CRP for each subject by cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Lasseter, MD, Principal Investigator — Clinical Pharmacology of Miami; Richard Straube, MD, Study Director — Stealth BioTherapeutics Inc.
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States